CLINICAL TRIAL: NCT03111810
Title: Targeting Iatrogenic Cushing's Syndrome With 11β-hydroxysteroid Dehydrogenase Type 1 Inhibition (TICSI)
Brief Title: Targeting Iatrogenic Cushing's Syndrome With 11β-hydroxysteroid Dehydrogenase Type 1 Inhibition
Acronym: TICSI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 212634
Record Dates: First submitted 2017-03-17; First posted 2017-04-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-03

CONDITIONS: Iatrogenic Cushing's Disease
Keywords: Corticosteroids; Prednisolone; 11 beta-Hydroxysteroid dehydrogenase1 inhibitor; Iatrogenic Cushing's disease; AZD4017
MeSH Terms: interventions — 2-(1-(5-(cyclohexylcarbamoyl)-6-propylsulfanylpyridin-2-yl)-3-piperidyl)acetic acid; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): Prednisolone 20mg once daily and AZD4017 400mg twice daily for 7 days.
  Interventions: Drug: AZD4017 and prednisolone
- Placebo Oral Tablet (Placebo Comparator): Prednisolone 20mg once daily and placebo twice daily for 7 days.
  Interventions: Drug: Placebo Oral Tablet and prednisolone

INTERVENTIONS:
Drug: AZD4017 and prednisolone — The drug AZD4017 will be given together with prednisolone 20mg daily for 7 days to compare its effects on metabolic tissues against the placebo arm where the participants will take placebo and prednisolone 20mg daily for 7 days.
  Other Names: 11 beta-Hydroxysteroid dehydrogenase inhibitor
  Arms: Active
Drug: Placebo Oral Tablet and prednisolone — Placebo Oral tablet will be given together with prednisolone 20mg daily for 7 days to compare the effects on metabolic tissues of AZD4017 and prednisolone 20mg daily against the placebo arm.
  Other Names: Placebo
  Arms: Placebo Oral Tablet

SUMMARY:
Currently, 2-3% of the population of the United Kingdom and United States of America receive glucocorticoid therapy. Significant adverse effects are not confined to chronic use; recurrent short-course administration is associated with increased morbidity and mortality. The adverse metabolic features associated with glucocorticoid use include obesity, skeletal muscle myopathy, hypertension, insulin resistance and diabetes and are collectively termed 'iatrogenic Cushing's syndrome'. The efficacy of glucocorticoid therapy is not in doubt, but there are no interventions to reduce their metabolic consequences. Within metabolic tissues (liver, skeletal muscle, adipose), 11β-hydroxysteroid dehydrogenase type 1 (11β-HSD1) regenerates active glucocorticoid and therefore is able to tightly control the availability of glucocorticoids to activate the glucocorticoid receptor. In preclinical studies, the investigators have shown that 11β-HSD1 is critical in regulating the development of the adverse features associated with circulating glucocorticoid excess, endorsing our observations in a patient with Cushing's disease, who was protected from a classical phenotype due to a functional deficit in 11β-HSD1.

This study is the first clinical evaluation of the impact of the selective 11β-HSD1 inhibitor, AZD4017, in healthy volunteers taking exogenous glucocorticoids (prednisolone). The investigators propose that in tissues expressing high levels of 11β-HSD1, prednisolone action will be amplified, driving adverse effects within these tissues and have hypothesized that AZD4017 in humans will reduce the adverse metabolic consequences of Prednisolone administration without compromise to its anti-inflammatory action.

Our specific research objectives are:

1. To demonstrate the beneficial effect of the selective 11β-HSD1 inhibitor, AZD4017, upon the prednisolone-induced deterioration in metabolic phenotype, including glucose disposal and endogenous glucose production rates.
2. To determine the impact of AZD4017 on the anti-inflammatory actions of Prednisolone.
3. To identify the tissue-specific (skeletal muscle, adipose) mechanisms underpinning the response to Prednisolone therapy administered in conjunction with AZD4017.

The investigators will perform a randomized, double-blind placebo controlled study to determine if co-administration of the selective 11β-HSD1 inhibitor, AZD4017, limits the adverse effects of short-course exogenous glucocorticoid administration. 32 healthy male volunteers will have detailed metabolic investigations including 2-step hyperinsulinaemic euglycaemic clamps (with stable isotope measurements of lipid and carbohydrate metabolism), as well as assessment of skeletal muscle forearm glucose uptake. All volunteers will then be treated with Prednisolone (20mg daily) and randomized to the co-administration of placebo or AZD4017. After 1 week of therapy, all investigations will be repeated. Our hypothesis is that the adverse metabolic effects of Prednisolone will be reduced by co-administration of AZD4017.

ELIGIBILITY:
Inclusion Criteria:

The following criteria apply to both arms and each volunteer who has a successful screening visit will be randomized to one of the arms defined above (see section 6): We estimate that we will need to screen 40-50 patients in order to achieve our recruitment target.

* Male volunteers without diabetes (HbA1C < 48mmol/mol at screening)
* BMI 20-30kg/m2
* Age 18-60years
* For individuals identified from Oxford Biobank - fasting insulin and / or glucose and / or insulin resistance as measured by Homeostatic model assessment (HOMA) - insulin resistance in the 40th-60th percentile
* BP<160/100 mmHg with stable antihypertensive therapy for >3 months
* Stable lipid lowering therapy for >3 months
* No contraindications to AZD4017 or prednisolone treatment Study participants who are sexually active with a female partner of childbearing potential must be surgically sterilized, practicing true abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence, e.g. calendar, ovulation, symptothermal, post-ovulation methods, declaration of abstinence for the duration of a trial, and withdrawal are not acceptable methods of contraception) or agree, along with their partners, to use two forms of highly effective methods of birth control (i.e. condom plus another highly effective method defined below), and not rely on barrier methods and spermicide alone, from the time of screening and for the duration of the study. For the proposed clinical study, all study subjects will be male.

For male study subjects whose partner is pregnant, or whose partner is a woman of child-bearing potential (WOCBP) who is established on and continuing to use a highly effective method of contraception, in addition to the stipulations above, males should continue to use a condom (in addition to the highly effective method) for 1 week following the last dose of study drug (5 drug elimination half-lives rounded up to 1 week).

For male study subjects whose partner is not pregnant but is a WOCBP who is not established on and continuing to use a highly effective method of contraception, males should continue to use a condom (in addition to the highly effective method) for 3 weeks following the last dose of study drug (5 drug elimination half-lives plus 2 weeks).

Male study participants must also not donate sperm from the time of screening until 3 weeks after final dose of study drug (5 drug elimination half-lives plus 2 weeks).

Highly effective methods of contraception are defined as combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (either oral, intravaginal or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (either oral [specifically Cerazette™], injectable or implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner or sexual abstinence.

We would advise that competitive elite athletes do not take part in the study as there is the possibility that the prednisolone could impact upon their athletic performance

Exclusion Criteria:

The participant may not enter the study if any of the following apply:

* Age <18 or >60years
* Body mass index <20 or >30kg/m2
* A diagnosis of diabetes (type 1 or type 2)
* A blood haemoglobin <120mg/dL
* Haemorrhagic disorders
* Anticoagulant treatment
* Renal impairment with estimated Glomerular Filtration Rate <60ml/min
* Abnormal liver chemistry with aspartate aminotransferase, alanine transaminase and/or Gamma-glutamyltransferase and/or bilirubin more than the upper limit of normal
* Glucocorticoid therapy (including inhaled, topical or oral) within the last 6 months
* Concomitant anti-inflammatory medication including NSAIDs, disease modifying anti-rheumatic drugs (DMARDs) / steroid-sparing medications (e.g. methotrexate, sulphasalazine, hydroxychloroquine, azathioprine, leflunomide, biologics [anti-Tumor necrosis factor alpha, interleukin-1ra]).
* Any medical condition in the opinion of the investigator that might impact upon safety or validity of the results - recent (within 2 weeks) or active infection, known liver disease, known thyroid disease, active malignancy, existing inflammatory condition (e.g. inflammatory arthropathy, inflammatory bowel disease, autoimmune disease, connective tissue disease)
* Current evidence of alcohol abuse or a significant history of alcohol abuse, as judged by the investigator.
* Contraindication to any of the study treatments or known or suspected hypersensitivity to the investigational product, compounds of the same class, other study treatments or any excipients.
* Unwilling, or unable, to give informed consent.
* Participation in another investigational medicinal product trial / study within the past 6 months

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Changes in the detrimental side effects of prednisolone by AZD4017. | 2 years
  To evaluate whether AZD4017 can limit the detrimental effect of prednisolone (20mg) on glucose disposal. This will be achieved by measuring glucose disposal during a hyperinsulinaemic euglycaemic clamp.

SECONDARY OUTCOMES:
Changes in hepatic insulin sensitivity by AZD4017 when given with prednisolone (20mg) compared to prednisolone (20mg) given alone. | 2 years
  Measurement of endogenous glucose production rate during a hyperinsulinaemic euglycaemic clamp.
Changes in blood pressure associated with prednisolone and AZD4017 administration | 2 years
  The participants will have 24h ambulatory blood pressure measurements taken.
Changes in adipose tissue gene expression profile associated with prednisolone and AZD4017 administration. | 2 years
  Gene expression changes will be measured from adipose tissue biopsies.
Change in whole body oxidation associated with prednisolone and AZD4017 administration | 2 years
  Measurement of incorporation of carbon-13 into breath carbon dioxide using Gas chromatography combustion isotope ratio mass spectrometry.
Changes in skeletal muscle gene expression profile associated with prednisolone and AZD4017 administration. | 2 years
  Gene expression changes measured in skeletal muscle biopsies.
Changes in circulating inflammatory cytokines and inflammatory response in circulating inflammatory cells associated with prednisolone and AZD4017 administration. | 2 years
  Measurement of inflammatory cytokines, isolation of peripheral blood mononuclear cells and defining their response to inflammatory stress.
Changes in bone turnover associated with prednisolone and AZD4017 administration. | 2 years
  Measurement of serum and urine markers of bone turnover including type I collagen cross-linked N-telopeptide and osteocalcin
Changes in body composition (total and regional lean and fat mass) associated with prednisolone and AZD4017 administration. | 2 years
  Measurement of total and regional lean and fat mass on dual energy x-ray absorptiometry scan.
Changes in urinary steroid metabolite profile associated with prednisolone and AZD4017 administration. | 2 years
  Steroid metabolites measured by gas chromatography, mass spectrometry in a timed overnight urine sample.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Staa TP, Leufkens HG, Abenhaim L, Begaud B, Zhang B, Cooper C. Use of oral corticosteroids in the United Kingdom. QJM. 2000 Feb;93(2):105-11. doi: 10.1093/qjmed/93.2.105. PMID 10700481
- [Background] Overman RA, Yeh JY, Deal CL. Prevalence of oral glucocorticoid usage in the United States: a general population perspective. Arthritis Care Res (Hoboken). 2013 Feb;65(2):294-8. doi: 10.1002/acr.21796. PMID 22807233
- [Background] Gathercole LL, Lavery GG, Morgan SA, Cooper MS, Sinclair AJ, Tomlinson JW, Stewart PM. 11beta-Hydroxysteroid dehydrogenase 1: translational and therapeutic aspects. Endocr Rev. 2013 Aug;34(4):525-55. doi: 10.1210/er.2012-1050. Epub 2013 Apr 23. PMID 23612224
- [Background] Morgan SA, McCabe EL, Gathercole LL, Hassan-Smith ZK, Larner DP, Bujalska IJ, Stewart PM, Tomlinson JW, Lavery GG. 11beta-HSD1 is the major regulator of the tissue-specific effects of circulating glucocorticoid excess. Proc Natl Acad Sci U S A. 2014 Jun 17;111(24):E2482-91. doi: 10.1073/pnas.1323681111. Epub 2014 Jun 2. PMID 24889609
- [Background] Tomlinson JW, Draper N, Mackie J, Johnson AP, Holder G, Wood P, Stewart PM. Absence of Cushingoid phenotype in a patient with Cushing's disease due to defective cortisone to cortisol conversion. J Clin Endocrinol Metab. 2002 Jan;87(1):57-62. doi: 10.1210/jcem.87.1.8189. PMID 11788623
- [Background] Scott JS, Bowker SS, Deschoolmeester J, Gerhardt S, Hargreaves D, Kilgour E, Lloyd A, Mayers RM, McCoull W, Newcombe NJ, Ogg D, Packer MJ, Rees A, Revill J, Schofield P, Selmi N, Swales JG, Whittamore PR. Discovery of a potent, selective, and orally bioavailable acidic 11beta-hydroxysteroid dehydrogenase type 1 (11beta-HSD1) inhibitor: discovery of 2-[(3S)-1-[5-(cyclohexylcarbamoyl)-6-propylsulfanylpyridin-2-yl]-3-piperidyl]acetic acid (AZD4017). J Med Chem. 2012 Jun 28;55(12):5951-64. doi: 10.1021/jm300592r. Epub 2012 Jun 19. PMID 22691057
- [Background] Hazlehurst JM, Gathercole LL, Nasiri M, Armstrong MJ, Borrows S, Yu J, Wagenmakers AJ, Stewart PM, Tomlinson JW. Glucocorticoids fail to cause insulin resistance in human subcutaneous adipose tissue in vivo. J Clin Endocrinol Metab. 2013 Apr;98(4):1631-40. doi: 10.1210/jc.2012-3523. Epub 2013 Feb 20. PMID 23426618
- [Background] Tripathy D, Daniele G, Fiorentino TV, Perez-Cadena Z, Chavez-Velasquez A, Kamath S, Fanti P, Jenkinson C, Andreozzi F, Federici M, Gastaldelli A, Defronzo RA, Folli F. Pioglitazone improves glucose metabolism and modulates skeletal muscle TIMP-3-TACE dyad in type 2 diabetes mellitus: a randomised, double-blind, placebo-controlled, mechanistic study. Diabetologia. 2013 Oct;56(10):2153-63. doi: 10.1007/s00125-013-2976-z. Epub 2013 Jun 30. PMID 23811853
- [Derived] Gomez C, Alimajstorovic Z, Othonos N, Winter DV, White S, Lavery GG, Tomlinson JW, Sinclair AJ, Odermatt A. Identification of a human blood biomarker of pharmacological 11beta-hydroxysteroid dehydrogenase 1 inhibition. Br J Pharmacol. 2024 Mar;181(5):698-711. doi: 10.1111/bph.16251. Epub 2023 Oct 19. PMID 37740611